CLINICAL TRIAL: NCT07141407
Title: Community-Engaged Pilot Testing of Talking About Cancer (TAC) to Improve Engagement in Advance Care Planning
Brief Title: Telephone-Based Coaching Sessions (TAC) to Improve Advance Care Planning Participation in Advanced Cancer Patients and Their Support Person
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fred Hutchinson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: RG1125666; NCI-2025-05520 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); FHIRB0020936 (Other: Fred Hutch/University of Washington Cancer Consortium)
Record Dates: First submitted 2025-08-19; First posted 2025-08-26 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Advanced Malignant Solid Neoplasm; Hematopoietic and Lymphatic System Neoplasm
MeSH Terms: interventions — Palliative Care; Early Intervention, Educational; Educational Status; Methods

STUDY DESIGN:
Who Masked: Care Provider
Masking Description: The study project coordinator will oversee randomization and the research coordinator conducting assessments will remain blind to the condition to which the participant is assigned.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm I (TAC sessions) (Experimental): Participants attend Talking About Cancer (TAC) telephone-based coaching sessions (2 sessions) designed to support participants in communicating about advance care planning (ACP), managing distress around ACP conversations, engaging in the process of ACP, and completing advance directives over 45-60 minutes each once a week (QW) for 2 weeks.
  Interventions: Other: Supportive Care; Behavioral: Telephone-Based Intervention; Other: Survey Administration
- Arm II (enhanced usual care) (Active Comparator): Participants receive an ACP brochure/handout on study.
  Interventions: Other: Survey Administration; Other: Educational Intervention

INTERVENTIONS:
Other: Supportive Care — Attend TAC telephone-based coaching sessions
  Other Names: Supportive Therapy; Symptom Management; Therapy, Supportive
  Arms: Arm I (TAC sessions)
Behavioral: Telephone-Based Intervention — Attend TAC telephone-based coaching sessions
  Arms: Arm I (TAC sessions)
Other: Survey Administration — Ancillary studies
Other: Educational Intervention — Receive an ACP brochure/handout
  Other Names: Education for Intervention; Intervention by Education; Intervention through Education; Intervention, Educational
  Arms: Arm II (enhanced usual care)

SUMMARY:
This clinical trial studies whether telephone-based coaching sessions, Talking About Cancer (TAC), work to improve engagement in advance care planning (ACP) in patients with cancer that may have spread from where it first started to nearby tissue, lymph nodes, or distant parts of the body (advanced) and their support person. Participation in ACP, which includes having end of life (EOL) care conversations and completing advance directives (e.g., living will, health care proxy, do not resuscitate order), improves quality EOL care. Despite this, less than half of patients with advanced cancer have EOL care conversations or complete advance directives. TAC coaching sessions are delivered by a social worker over the phone. They are designed to help patients and their support person communicate about ACP, manage the distress these conversations can cause, and participate in the process of ACP with a clear action plan of having goals-of-care conversations and completing advance directives. This may be an effective way to improve ACP participation in advanced cancer patients and their support person.

DETAILED DESCRIPTION:
OUTLINE: Participants are randomized to 1 of 2 arms.

ARM I: Participants attend Talking About Cancer (TAC) telephone-based coaching sessions (2 sessions) designed to support participants in communicating about advance care planning (ACP), managing distress around ACP conversations, engaging in the process of ACP, and completing advance directives over 45-60 minutes each once a week (QW) for 2 weeks.

ARM II: Participants receive an ACP brochure/handout on study.

After completion of study intervention, participants are followed up at 6- and 12-weeks post-randomization.

ELIGIBILITY:
Inclusion Criteria:

* PATIENT: Current diagnosis of stage III or IV cancer
* PATIENT: Able to provide informed consent
* PATIENT: Fluent in English or Spanish
* PATIENT: Have access to a telephone, computer, or mobile device
* CAREGIVER (SUPPORT PERSON): Person patient indicates provides support
* CAREGIVER (SUPPORT PERSON): English or Spanish speaking
* CAREGIVER (SUPPORT PERSON): 18 years of age or older
* CAREGIVER (SUPPORT PERSON): Able to provide informed consent

Exclusion Criteria:

* PATIENT: Too ill or weak to complete the interviews (as judged by the interviewer)
* PATIENT: Receiving hospice at the time of enrollment
* PATIENT: Younger than age 18

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2026-04-01 (Estimated); Primary Completion 2026-10-12 (Estimated); Study Completion 2026-12-14 (Estimated)

PRIMARY OUTCOMES:
Enrollment rate (Feasibility) | At 6-weeks post-randomization
  Feasibility will be examined using enrollment rates. Feasibility cutoffs will be based on prior research and include the following: ≥ 50% of eligible participants will enroll in the study. Low rates of enrollment, including missing data, will indicate low feasibility.
Intervention session completion rate (Feasibility) | At 6-weeks post-randomization
  Feasibility will be examined using enrollment and intervention completion rates as outcomes. Feasibility cutoffs will be based on prior research and include the following: ≥ 75% of Talking About Cancer sessions will be delivered with fidelity.
Acceptability of Intervention Measure (AIM) score (Acceptability) | At 6-weeks post-randomization
  To analyze intervention acceptability, will examine the median score for the AIM measure, with a median of >= 4 indicating acceptability (on a 5-point Likert scale where 4=Agree and 5=Completely agree and higher scores indicate higher levels of acceptability).
Completion rate of study assessments (Feasibility of collecting primary and secondary outcomes) | At baseline, 6-weeks post- randomization, and 12-weeks post-randomization
  Feasibility of the study collection procedures will be examined using study-related assessment completion rates and includes the following: ≥ 50% of enrolled patients will adhere to and complete assigned intervention components and study-related assessments.

SECONDARY OUTCOMES:
Completion of advance directives | At baseline, 6-weeks post-randomization, and 12-weeks post-randomization
  Completion of advance directives will be assessed with questions that ask patients (caregivers) whether the patient has completed a do not resuscitate (DNR) order, living will or identified a health care proxy. This item is scored as having not advance directives (0) to all advance directives completed (3). In addition to the primary outcome of advance directives (0 to 3 score), will also examine each outcome separately (e.g., yes/no to completing a health care proxy) as secondary measures. Descriptive statistics will be run, including means and standard deviations for continuous data and frequencies and proportions for categorical data. Bivariate correlations will be run between demographics and clinical characteristics to determine if any are associated with the primary outcome at baseline.
Completion of do not resuscitate (DNR) order | At baseline, 6-weeks post-randomization, 12-weeks post-randomization
  Completion of advance directives will be assessed with questions that ask patients (caregivers) whether the patient has completed a DNR order. This item is scored as having not advance directives (0) to all advance directives completed (3). In addition to the primary outcome of advance directives (0 to 3 score), will also examine each outcome separately (e.g., yes/no to completing a health care proxy) as secondary measures. Descriptive statistics will be run, including means and standard deviations for continuous data and frequencies and proportions for categorical data.
Completion of living will | At baseline, 6-weeks post-randomization, and 12-weeks randomization
  Completion of advance directives will be assessed with questions that ask patients (caregivers) whether the patient has completed a living will. This item is scored as having not advance directives (0) to all advance directives completed (3). In addition to the primary outcome of advance directives (0 to 3 score), will also examine each outcome separately (e.g., yes/no to completing a health care proxy) as secondary measures. Descriptive statistics will be run, including means and standard deviations for continuous data and frequencies and proportions for categorical data.
Identification of a health care proxy | At baseline, 6-weeks post-randomization, and 12-weeks post-randomization
  Completion of advance directives will be assessed with questions that ask patients (caregivers) whether the patient has identified a health care proxy. This item is scored as having not advance directives (0) to all advance directives completed (3). In addition to the primary outcome of advance directives (0 to 3 score), will also examine each outcome separately (e.g., yes/no to completing a health care proxy) as secondary measures. Descriptive statistics will be run, including means and standard deviations for continuous data and frequencies and proportions for categorical data.
Advance care planning (ACP) conversations | At baseline, 6-weeks post-randomization, and 12-weeks post-randomization
  Will be assessed with the previously utilized 8-item measure of discussing end-of-life care (e.g., goals of care conversation), living will, health care proxy and DNR orders with doctor(s) and family members/loved ones. Descriptive statistics will be run, including means and standard deviations for continuous data and frequencies and proportions for categorical data.
Level of engagement in ACP | At baseline, 6-weeks post-randomization, and 12-weeks post-randomization
  Will be measured using the reliable and valid Advance Care Planning Engagement Survey: Action Measures. It is an 18-item measure assessing domains of decision maker, quality of life, flexibility, and asking questions about treatment and ACP (yes/no). Descriptive statistics will be run, including means and standard deviations for continuous data and frequencies and proportions for categorical data.
Readiness to engage in ACP | At baseline, 6-weeks post-randomization, and 12-weeks post-randomization
  Will be assessed using the previously developed and validated questionnaire, the Advance Care Planning Readiness Scale. This is an 8-item questionnaire that asks questions about patients' readiness to engage in ACP on a 7-point Likert scale (1=Strongly disagree, 7 = Strongly agree). Descriptive statistics will be run, including means and standard deviations for continuous data and frequencies and proportions for categorical data.
Self-efficacy for treatment decision-making | At baseline, 6-weeks post-randomization, and 12-weeks post-randomization
  Will be measured by the Decision-Making Participation Self-Efficacy (DEPS) scale. The DEPS scale is a 5-item validated measure that assesses cancer patients' confidence in engaging in different activities related to decision-making. Patients are asked to indicate how confident they are that they would be able to engage in various decision-making activities (e.g., "Tell your doctor about the option you would prefer"); items are rated on a 5-point Likert scale (0 = not at all confident, 4 = completely confident). Descriptive statistics will be run, including means and standard deviations for continuous data and frequencies and proportions for categorical data.
Psychological distress | At baseline, 6-weeks post-randomization, and 12-weeks post-randomization
  Will be measured using the Hospital Anxiety and Depression Scale, a valid and reliable 14-item, Likert-type self-report measure of mood disturbance commonly used with cancer patients. Descriptive statistics will be run, including means and standard deviations for continuous data and frequencies and proportions for categorical data.
Prognostic understanding | At baseline, 6-weeks post-randomization, and 12-weeks post-randomization
  Will be assessed with items used previously in the team's National Institutes of Health-funded cohort studies of advanced cancer patients and their caregivers: terminal nature of the illness (terminal [accurate] versus non-terminal [inaccurate]) and life-expectancy (months [accurate] versus years [inaccurate]). Descriptive statistics will be run, including means and standard deviations for continuous data and frequencies and proportions for categorical data.
Support person [caregiver] burden | At baseline, 6-weeks post-randomization, and 12-weeks post-randomization
  Will be measured using the Zarit Burden Interview, a reliable and valid 22-item measure of caregiver burden used in intervention studies of cancer caregivers. Descriptive statistics will be run, including means and standard deviations for continuous data and frequencies and proportions for categorical data.

CONTACTS AND LOCATIONS:
Overall Officials: Megan Shen, PhD, Principal Investigator — Fred Hutch/University of Washington Cancer Consortium
Locations (1):
- Fred Hutch/University of Washington Cancer Consortium, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No